CLINICAL TRIAL: NCT04258124
Title: Effectiveness of a Physical Therapy Intervention Through Cervical Motor Control Exercises in the Improvement of Strength and Perception of Effort in Electronic Sports Players. A Randomized Clinical Study
Brief Title: Cervical Motor Control Exercises in Strength and Perception of Effort in Electronic Sports Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMOTOR
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Sports Physical Therapy
Keywords: Physiotherapy; Motor Control; Cervical; Stabilizer; Esports

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 10 minutes, taking place 3 days a week, over a period of 6 weeks. The intervention will take place at the beginning of the training session. The intervention will be carried out in 3 sessions with 3 exercises of 15 repetitions, and with breaks of 40 seconds between each series and exercise.
  Exercise 1. In quadruped position, keeping the back flat, making an isometric contraction of the transverse muscle, and raising one arm and one leg contralaterally.
  Exercise 2. Training of the deep cervical flexor muscles, supine. Players will move their heads slowly towards craniocervical flexion.
  Exercise 3. In standing position, an ocular-cervical coordination exercise by means of a cranio-cervical flexion, adding a rotation, guided by an eye feedback provided by the physiotherapist by means of a laser projected on a wall.
  Interventions: Other: Control motor intervention
- Control group (No Intervention): Athletes in the control group will be asked to follow their usual warm-up routine.

INTERVENTIONS:
Other: Control motor intervention — The intervention through motor control will consist in the application of the protocol described by Hidalgo-Peréz et al. The objective of the application of the technique is to produce an increase in the strength of the deep cervical musculature. The exercises will be performed with the subject in different positions: supine, quadrupedic and standing position. The physiotherapist will be placed in standing position in front of the subject. The intervention will be carried out in 3 sessions with 3 exercises of 15 repetitions, and with breaks of 40 seconds between each series and exercise.
  Arms: Experimental group

SUMMARY:
Introduction. One of the most common injuries in competitive esports professionals is dorsolumbar and neck pain, due to the effort caused by the maintenance of the site for long periods of time. Cervical motor control exercises recruit the deep musculature by increasing its strength and reducing muscle fatigue.

Aim. Evaluate the effectiveness of motor control exercises in cervical muscle fatigue and strength, in electronic athletes from 18 to 25 years.

Study design. Randomized clinical trial, simple blind. Methods. 30 electronic athletes will be randomly assigned in two groups: experimental (which will perform 3 sessions of 3 motor control exercises) and control (which will not perform any type of intervention). The intervention will last 6 weeks, with 3 weekly sessions of 10 minutes each. The study variables are the muscle strength of the deep cervical muscle (measured by a stabilizer pressure gauge) and the subjective perception of the effort (Borg scale).

Expected results. The aim is an improvement in the muscular strength of deep cervical muscles, together with a decrease in subjective perception of exertion.

ELIGIBILITY:
Inclusion Criteria:

* Electronic sportsmen
* Male sex
* From 18 to 25 years
* That at the time of the study participate in national competitions
* That they have not suffered a musculoskeletal pathology in the last 4 months.

Exclusion Criteria:

* Athletes taking anti-inflammatory drugs that may influence the intervention
* Players who are allergic to nylon (main component of the evaluation device)
* That they have not signed the informed consent document.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-24 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline strength of the deep cervical musculature after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An assessment will be carried out with a pressure gauge (Stabilizer model). It will be used according to the protocol indicated by Hudswell et al. The athlete will be positioned supine. The pressure gauge will be placed on the stretcher in the posterior cervical area, asking the subject for a craniocervical flexion. The unit of measure of this measuring instrument is mmHg. A higher score indicates greater strength.

SECONDARY OUTCOMES:
Change from baseline subjective perception of effort after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by administering the Borg scale. With this scale, the perception of effort will be measured. After the intervention, we will ask the athlete to assign a number from 0 to 10 to represent the subjective feeling of the amount of work done. The scoring range is from 0 to 10 points, where a higher score will indicate a greater perception of effort.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- European University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided